CLINICAL TRIAL: NCT05584488
Title: Natural History Study for Genetic Diseases of Allergic Inflammation and Immune Dysregulation
Brief Title: Allergy and Immunology Natural History Study
Status: Recruiting | Type: Observational
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Other Study IDs: AAAS7006
Record Dates: First submitted 2022-10-14; First posted 2022-10-18 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Immune Deficiency; Immune Dysregulation Disorder; Allergic Inflammation
Keywords: Eosinophilic Disease; Anaphylaxis; Elevated IgE levels; Autoimmune diseases; Allergy; Asthma; Atopic Dermatitis; Allergic Fhinitis; Food Allergy; Immunodeficiency Diseases; Immunodysregulatory Diseases; Piebaldism; Urticaria; Angioedema
MeSH Terms: conditions — Immunologic Deficiency Syndromes; Anaphylaxis; Autoimmune Diseases; Hypersensitivity; Asthma; Dermatitis, Atopic; Food Hypersensitivity; Piebaldism; Urticaria; Angioedema

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood specimens, stored blood samples, stored blood products (including cells, DNA, RNA, and protein), saliva, hair, finger nail clippings, cord blood, umbilical cord, tissue biopsy, bone marrow and/or buccal swabs will be obtained from patients and/or their blood relatives.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Inherited diseases of allergic inflammation or immune dysregulation: Patients and blood relatives with disorders of allergic inflammation and immune dysregulation.

SUMMARY:
This protocol is a natural history study designed to evaluate subjects (and some family members) with suspected or identified genetic diseases of allergic inflammation or Immune Dysregulation. Patients determined by clinical history and outside evaluations to be of interest will be consented and enrolled into this study. Blood specimens, stored blood products and derivatives, saliva, hair, fingernail clippings, cord blood, umbilical cord, bone marrow, tissue biopsies and/or buccal swabs from such patients and/or their family members will be obtained for research studies related to understanding genetic and immunopathogenic bases of these diseases. Outside medical records may be obtained, and patient evaluations may be performed to correlate to research laboratory testing results.

DETAILED DESCRIPTION:
Studying patients with suspected genetic diseases with features of atopy or affecting atopic pathways, both known and novel disorders, will provide critical populations for understanding atopic pathways and mechanisms of allergic inflammation in atopic dermatitis, and atopic diseases in general. This investigation will include patients with atopic diseases and other related syndromes and both their healthy and ill family members. The goal of these studies is to advance understanding of the genetic and immunologic basis of disorders of allergic inflammation, leading to the development of improved methods for the diagnosis and management of patients with atopic diseases, immunodeficiency, and immune dysregulatory diseases. Immune dysregulation diseases comprise a group of disorders that can trigger defective or uncontrolled immune responses and are characterized by autoimmunity, episodes of recurrent autoinflammation, dysregulation of lymphocyte homeostasis, or hypersensitivity reactions. In addition to classical atopy, the investigators also use this line of research to further study other abnormalities affecting immune dysregulation. Patients with idiopathic anaphylaxis are also of interest.

The continued dissection of the genetic and biochemical bases of known and, as yet, undiscovered defects will have an impact beyond the mast cell and will contribute to the development of new therapies. This investigation will include patients with these and other related syndromes and both their healthy and ill family members. Moreover, these studies will continue to provide a wealth of information about the regulation of allergy and mast cell homeostasis in normal individuals. Research into these fundamental processes will help provide an understanding of how conditions of immediate hypersensitivity and cancers generally arise, and could lead to new preventative measures, diagnostic tests, treatments, or cures for these conditions.

The investigators propose to evaluate subjects who may have, or are suspected of having, inherited diseases of allergic inflammation or Immune Dysregulation which may include the following diseases:

* Autoimmune diseases
* Anaphylaxis
* Allergy
* Asthma
* Atopic dermatitis
* Allergic rhinitis
* Food allergy
* Immunodeficiency diseases
* Immunodysregulatory diseases
* Piebaldism
* Urticaria/angioedema

ELIGIBILITY:
Inclusion Criteria:

* Subjects, ages birth to 99 years old, known to have or suspected of having an inherited disorder of allergic inflammation, or mast cell homeostasis, or activation or immune dysregulation.
* Blood relatives of enrolled subjects will be eligible for enrollment.
* There will be no discrimination as to age, gender, race, or disability.
* Subjects/guardians must be willing and able to give informed consent.
* Subjects must agree to have their blood stored for future studies of the immune system and/or other medical conditions.

Exclusion Criteria:

• The presence of an acquired abnormality of the immune system, such as cytotoxic chemotherapy or malignancy may be grounds for possible exclusion if, in the opinion of the investigator, the presence of such a disease process would interfere with evaluation.

Max Age: 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The total study population for this protocol is up to 10,000 subjects. It is estimated that one half of the total study population will consist of subjects, with the remaining half being biological relatives. Subjects and relatives may be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2010-07-16 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Total number of underlying susceptibility trait(s) identified | Up to 1 year
  The primary endpoint will be the determination of the underlying susceptibility trait(s).

CONTACTS AND LOCATIONS:
Overall Officials: Joshua D. Milner, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center / NewYork-Presbyterian Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No